CLINICAL TRIAL: NCT04110327
Title: An All-Comers Observational Study of the MicroStent™ Peripheral Vascular Stent System in Subjects With Peripheral Arterial Disease
Acronym: HEAL
Status: Active, not recruiting | Type: Observational
Sponsor: Micro Medical Solution, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MMS-201
Record Dates: First submitted 2019-09-27; First posted 2019-10-01 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2024-12

CONDITIONS: Peripheral Arterial Disease; Critical Lower Limb Ischemia
Keywords: MicroStent; Below the Knee; CLI; Below the Ankle; CLTI
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: MicroStent — Treatment of arterial stenosis or occlusion with the MicroStent Peripheral Vascular Stent System

SUMMARY:
Non-randomized, multicenter, combined prospective and retrospective cohort analysis consisting of a single arm treated with the MicroStent™ System.

DETAILED DESCRIPTION:
Subjects with peripheral arterial disease (PAD) whom the investigator has treated or intends to treat with the MicroStent™ System per the current instructions for use (IFU), and who have given written informed consent, will be enrolled in this study. Up to 300 subjects will be enrolled:

The objective of this post market registry is to evaluate procedural and long-term clinical outcomes for subjects undergoing intervention with the MicroStent® System for treatment of lower extremity peripheral arterial disease (PAD), presenting with below-the-knee lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Any subject with below the knee, at the ankle level or below the ankle peripheral arterial lesions previously treated or intended to be treated with the MicroStent® System per the current indications for use
2. For across the ankle joint intervention, distal runoff to digital branches or arcuate arteries must be present on angiography prior to MicroStent deployment
3. Subject's age is ≥ 18 years.
4. Subject must be willing to sign a patient informed consent form.

Exclusion Criteria:

1. Subject is pregnant or planning to become pregnant during the study duration
2. Subject has a life expectancy of less than one (1) year
3. Subject has a known allergy to concomitant medication, contrast agents (that cannot be medically managed), anti-platelet, anti-coagulant or thrombolytic medications
4. Subject is enrolled in another study that has not reached its primary endpoint at the time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include any subject with symptomatic peripheral arterial disease (PAD) that require intervention with the MicroStent™ System.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-10-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Patency | 6 months post-procedure
  Freedom from target lesion occlusion with no clinically driven target lesion revascularization (TLR)
Freedom from Perioperative Death and Major Adverse Limb Events (MALE) | 30 days post-procedure
  Freedom from all-cause death or major adverse limb events. Major adverse limb events include above-ankle amputation, new bypass graft or graft revision, and thrombectomy or thrombolysis involving the target lesion.

SECONDARY OUTCOMES:
Freedom from Major Adverse Limb Events | 6, 12, 24 Months
  Major adverse limb events include above-ankle amputation, new bypass graft or graft revision, and thrombectomy or thrombolysis involving the target lesion.
Freedom from Major Amputation | 6, 12, 24 Months
  Freedom from above-ankle amputation in the target limb
Freedom from Clinically Driven Target Lesion Revascularization (TLR) | 6, 12, 24 Months
  Freedom from any revascularization procedure with involvement of the target lesion that is due to complaints of leg pain or worsening leg pain, a progressing, non-healing ulcer, or new ulcer formation with or without the presence of an abnormal non-invasive test.
Wound Healing | 30 days, 6, 12, 24 Months
  Wounds will be identified at the baseline visit and classified as fully healed or not healed at each follow up visit.
Device Success | Procedure
  Operator assessment of successful device deployment and full coverage of the lesion as intended
Technical Success | Procedure
  Attainment of less than or equal to 30% residual stenosis by visual estimate in the treated lesion using only the study device according to the IFU (i.e. including post dilation at the discretion of the investigator)

CONTACTS AND LOCATIONS:
Locations (10):
- Univ.-Klinikum LKH Graz, Graz, Austria
- Belgium (3):
  - OLV Hospital, Aalst
  - A.Z. Sint-Blasius, Dendermonde
  - ZOL Genk, Genk
- Germany (3):
  - Klinikum Hochsauerland - Karolinen Hospital, Arnsberg
  - University Heart Center Freiburg - Bad Krozingen, Bad Krozingen
  - University of Leipzig, Leipzig
- Italy (2):
  - Policlinico Abano Terme, Abano Terme
  - Maria Cecilia Hospital, Cotignola
- St. Antonius Ziekenhuis, Nieuwegein, Netherlands

IPD SHARING:
Plan to Share IPD: No